CLINICAL TRIAL: NCT05883605
Title: Clinical Validation of the Wrist Blood Pressure Measuring Device Combei BP 880 W for Home Use According to "the Universal" Standard (AAMI/ESH/ISO)" in the General Population
Brief Title: Clinical Validation of The Combei BP 880 W
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Society for Vascular Health (Other)
Responsible Party: Principal Investigator, Catherine DOGNON HADDAD, Professor Roland Asmar, International Society for Vascular Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: VALCOMBW22
Record Dates: First submitted 2022-05-31; First posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Hypertension
Keywords: validation; Blood pressure.; wrist device; electronic BP device; home Blood pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- one population of normotensive and hypertensive (Other): treated and untreated normotensive and hypertensive patients
  Interventions: Device: Measuring blood pressure

INTERVENTIONS:
Device: Measuring blood pressure — Measuring blood pressure using electronic device and using a mercury sphygmomanometer

SUMMARY:
Clinical validation of the wrist blood pressure measuring device Combei BP 880 W for home use according to "the Universal Standard for the validation of blood pressure measuring devices by the Association for the Advancement of Medical Instrumentation/European Society of Hypertension/International Organization for Standardization (AAMI/ESH/ISO)" in the general population.

DETAILED DESCRIPTION:
Members of the AAMI, ESH and ISO committees achieved a consensus on an optimal validation standard and agreed on a single protocol for the validation of BP measuring devices that will replace all previous ones.

Therefore, the Association for the Advancement of Medical Instrumentation / European Society of Hypertension / International Organization for Standardization Universal Standard (AAMI/ESH/ISO 81060-2:2018) is now considered as the standard protocol for the validation of non-invasive blood pressure measuring device.

This study aims to demonstrate that the Combei BP 880 W wrist device fulfills the requirements of the new protocol of clinical validation and its Amendment 1, 2020-01 for limb circumference distribution criteria.

this is a monocentric, prospective, non-randomized, non-interventional, cross-study.

Combei BP 880 W wrist device (Sphygmomanometer Under Test, SUT). The reference device is the mercury sphygmomanometer The primary objective of the study is to assess the accuracy of the automatic oscillometric BP measuring device at the wrist level, the Combei BP 880 W, in the general population, following AAMI/ESH/ISO 81060-2:2018 protocol and its Amendment 1, 2020-01 for limb circumference distribution criteria.

The Combei BP 880 W device will pass the test if:

1. The differences of at least 255 individual paired determinations of the SUT and of the observers' readings with the reference sphygmomanometer for all subjects, calculated separately for systolic blood pressure and diastolic blood pressure, shall have the mean value of the differences, be within or equal to +/- 5.0mmHg and a standard deviation no greater than 8.0 mmHg.
2. For the systolic blood pressure and diastolic blood pressure of at least 85 subjects, the standard deviation of the averaged paired determinations per subject of the SUT and of the observers' readings with the reference sphygmomanometer shall meet the criteria listed in Table 1 of AAMI/ESH/ISO 81060-2:2018.

The secondary objective is to confirm the safety of use of this device, intended for home use.

Inclusion criteria

* Patient older than 12 years;
* Patient who signed the informed consent form;
* Patient followed-up at site (in-patient or out-patient);
* Patient with wrist circumference between 12.5 and 21.5 cm*. *in accordance with the Indications For Use of the Combei BP 880 W device.

Non-inclusion criteria

* Patient unable to give a consent or understand properly protocol information;
* Patient suffering from arrhythmia;
* Patient with poor quality of Korotkov sounds;
* Patient for whom K5 sounds are absent. The validation team will consist of three persons: two observers trained in accurate BP measurement and a supervisor.

  1. The reference sphygmomanometer is calibrated just before the beginning of the study.
  2. The observers are trained to the use of the SUT.
  3. In-patients or out-patients are included in the study after reading and signing the ICF.
  4. After inclusion, the patient is screened to verify that he/she satisfies the inclusion/non-inclusion criteria of the protocol. If not, the patient will be excluded from the study and no blood pressure measure will be performed on this patient.
  5. The patient is placed comfortably, and the reference sphygmomanometer is placed on his/her left upper arm, except if left upper arm is wounded. In this case, the reference sphygmomanometer is placed on his/her right upper arm.
  6. Measurements start with alternance between measurements with the reference sphygmomanometer and the SUT according to the same arm sequential BP measurements method.
  7. For each measurement with the reference sphygmomanometer, the two observers using mercury sphygmomanometers and a double-headed stethoscope, blinded from each other's result, and then by the supervisor using the tested device according to the manufacturer recommendations. The diastolic blood pressure should be measured at Korotkoff K5 sound. The agreement between the 2 observers will be checked all over the evaluation period by the supervisor to make sure that the difference between the two observers is no more than 4 mmHg for systolic and diastolic BP values.Otherwise, the measurement should be repeated. The intra individual BP variability for the reference BP measurements must be < 12 mmHg for SBP and < 8 mmHg for DBP.
  8. The results are written down on a source document and then reported in the CRF. Any AE, ADE or device malfunction occurring during the protocol will be also documented and reported in the CRF. For this study, all source documents should be written in English language.
  9. At the end of the measurements, the patient participation to the study is over.

Study procedures:

1. Validation team and pre-study training

   The validation team will consist of three persons: two observers trained in accurate BP measurement and a supervisor.

   The reference sphygmomanometer is calibrated just before the beginning of the study.

   The observers are trained to the use of the SUT.
2. Inclusion of the patients

   In-patients or out-patients of the investigational site are included in the study after reading and signing the ICF. After inclusion, the patient is screened to verify that he/she satisfies the inclusion/non-inclusion criteria of the protocol. If not, the patient will be excluded from the study and no blood pressure measure will be performed on this patient.
3. Cuffs

   The cuffs used for reference auscultatory BP measurement will have an inflatable bladder length that covers 75-100% of the arm circumference of each patient and width that covers 37-50% of the arm circumference.

   Detailed description of cuffs used for reference BP measurement will be reported for each patient.
4. Blood pressure measurements

The validation will be performed according to the (AAMI/ESH/ISO) Universal Standard validation protocol described in detail elsewhere10. The patients will have their reference BP measured by the two observers using a mercury sphygmomanometer and a double-headed stethoscope, blinded from each other's result, and then by the supervisor using the tested devices. The agreement between the 2 observers will be checked all over the evaluation period by the supervisor to make sure that the difference between the two observers is no more than 4 mmHg for systolic and diastolic BP values. Otherwise, the reference measurement should be repeated. The intra individual variability of the reference BP measurements must be < 12 mm Hg for SBP and < 8 mm Hg for DBP.

The circumference of the patient's upper arm will be measured to ensure that the cuff-size being used is adequate for the subject. The upper arm midpoint is first determined by marking the arm posteriorly at a point halfway between the acromion and olecranon, measured while the arm is flexed 90 degrees at the elbow with the palm facing up. The subject's upper arm circumference shall be determined by measuring at the midpoint of the upper arm while the elbow is relaxed, and the arm is dangling freely to the side.

The circumference of the patient's wrist will be measured to ensure that the circumference is within the acceptable range 12.5 - 21.5 cm for the Combei device, otherwise the subject will be excluded.

Measurements made by the mercury sphygmomanometer, will be performed according to the "same arm, consecutive measurements" (Figure 1), on the left arm supported at heart level.

Measurements by the Combei BP 880 W device will be performed at the wrist level of the same arm supported at the heart level, as recommended by the manufacturer with the following procedure.

1. Ask the subject to relax for 5-10 min.
2. make sure that the subject :

   * is comfortably seated with legs uncrossed and feet flat on the floor,
   * has the back, elbow and forearm supported,
   * has the measurement site at the level of the left ventricle of the heart,
   * and other conditions as recommended by the validation protocol and the device manual user.

In total, nine consecutive BP measurements will be performed in each patient using the mercury sphygmomanometers (5 times) and the tested devices (4 times).

All nine-sequential same-arm measurements will be recorded as shown in Table 2, starting with the standard mercury sphygmomanometer, followed by the device. A resting period of a minimum of 60 seconds shall be observed between the end of one measurement and the beginning of the following measurement.

Table 2: Sequential measurements of BP recorded by the standard mercury sphygmomanometer and the tested device:

R0 Entry BP, observers 1 and 2 each with the mercury standard T0 Device detection BP, supervisor R1 Observers 1 and 2 with mercury standard T1 Supervisor with the test instrument R2 Observers 1 and 2 with mercury standard T2 Supervisor with the test instrument R3 Observers 1 and 2 with mercury standard T3 Supervisor with the test instrument R4 Observers 1 and 2 with mercury standard

The first auscultatory and the first device measurement represent the recruitment pressures (R0 and T0) are not used in the evaluation of the test device accuracy. Each of the reference BP measurements (R) is the average of the simultaneous readings of the two observers. For each subject, the device measurements T1, T2 and T3 will be compared to observer measurements. Each of the test device measurements is compared to the average of the previous and succeeding reference BP readings (T1 vs average of R1 and R2, T2 vs average of R2 and R3, T3 vs average of R3 and R4).

At the end of the measurements, the patient participation to the study is over.

The Statistical Analysis: Differences are calculated by subtracting the reference BP measurement from the test device measurement. The mean BP difference (SUT versus reference sphygmomanometer) and its standard deviation (SD) will be calculated for the analysis. The same criteria will be used for systolic blood pressure and diastolic blood pressure measurements. The statistical analysis will be performed according to the requirements of the AAMI/ESH/ISO standard 2018 and its Amendment 1, 2020-01 for limb circumference distribution criteria.

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 12 years;
* Patient who signed the informed consent form;
* Patient followed-up at site (in-patient or out-patient);
* Patient with wrist circumference between 12.5 and 21.5 cm*. *in accordance with the Indications For Use of the Combei BP 880 W device.

Exclusion Criteria:

* Patient unable to give a consent or understand properly protocol information;
* Patient suffering from arrhythmia;
* Patient with poor quality of Korotkov sounds;
* Patient for whom K5 sounds are absent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Minimunn 30% male or female
Enrollment: 85 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2023-05-23 (Actual); Study Completion 2023-05-27 (Actual)

PRIMARY OUTCOMES:
Accuracy of blood pressure measurement | Subject will participate to only one session of measurement. The duration of one session is about 45 minutes.
  differences < than 5 +/- 8 mmHg according to the protocol by comparison to the gold standard (mercury sphygmomanometer)

SECONDARY OUTCOMES:
differences between the tested device and the gold standard (mercury sphygmomanometer according to the baseline blood pressure and to the wrist circumference | Subject will participate only one time to the study. one session of blood pressure measurement will be performed. the duration of one session is about 45 minutes
  differences < than 5 +/- 8 mmHg according to the protocol by comparison to the gold standard (mercury sphygmomanometer)

CONTACTS AND LOCATIONS:
Overall Officials: ROLAND ASMAR, Study Chair — International Society of Vascular Health
Locations (1):
- Roland Asmar, Paris, France